CLINICAL TRIAL: NCT03641560
Title: A Multicenter Phase 4, Open-label, Single-arm, Safety and Efficacy Study of Enzalutamide in Indian Patients With Progressive Metastatic Castration-Resistant Prostate Cancer (mCRPC) Previously Treated With Docetaxel-Based Chemotherapy
Brief Title: A Safety and Efficacy Study of Enzalutamide in Indian Patients With Progressive Metastatic Castration-Resistant Prostate Cancer (mCRPC) Previously Treated With Docetaxel-Based Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0413
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Progressive Metastatic Castration-Resistant Prostate Cancer (mCRPC); Enzalutamide; Xtandi; MDV3100
MeSH Terms: interventions — enzalutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Enzalutamide (Experimental): Participants with progressive mCRPC who had previously been treated with docetaxel-based chemotherapy received 160 milligrams (mg) (4 capsules of 40 mg) enzalutamide orally, once daily until disease progression, unacceptable toxicity or any other discontinuation criteria were met.
  Interventions: Drug: Enzalutamide; Drug: Androgen deprivation therapy (ADT)

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide was administered orally
  Other Names: MDV3100; Xtandi
Drug: Androgen deprivation therapy (ADT) — All participants were required to maintain ADT during study treatment, either using a Gonadotropin Releasing Hormone (GnRH) agonist/antagonist or having a history of bilateral orchiectomy

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability of enzalutamide in Indian patients with progressive mCRPC previously treated with docetaxel-based chemotherapy. This study also evaluated the effect of enzalutamide on prostate-specific antigen (PSA).

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation, signet cell or small cell histology.
* Subject with established diagnosis of metastatic castration-resistant prostate carcinoma.
* Subject is being newly initiated on Xtandi treatment (Enzalutamide).
* Subject has an estimated life expectancy of ≥ 6 months.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject who is not eligible to receive Xtandi as per the locally approved prescribing information.
* Subject participating or planning to participate in any interventional drug trial during the course of this trial.
* Subject has received investigational study within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject has any condition which makes the subject unsuitable for study participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (8):
- India (8):
  - Site IN00002, Ahmedabad
  - Site IN00004, Hubli
  - Site IN00008, Kolkata
  - Site IN00003, Nashik
  - Site IN00007, Nashik
  - Site IN00010, New Delhi
  - Site IN00001, Pune
  - Site IN00011, Surat

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/9785-CL-0413/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=26384&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Indian male participants with progressive mCRPC previously treated with docetaxel-based chemotherapy were enrolled in this study.
Pre-assignment Details: Eligible participants who met inclusion criteria and none of the exclusion criteria were enrolled.
Period: Overall Study
Arm/Group | Enzalutamide
Started | 52
Completed | 0
Not Completed | 52
Not completed — Withdrawal by Subject | 6
Not completed — Progressive disease | 40
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAF): The SAF consisted of all participants who took at least 1 dose of study drug, and was used for safety analyses.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 52
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment- Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavorable & unintended sign (including an abnormal laboratory finding [e.g. hematology, clinical chemistry, or urinalysis or other safety assessment e.g., ECGs, radiographic scans, vital signs measurements, physical examination]), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. TEAE was defined as an adverse event observed after starting administration of the study drug.
Time Frame: From first dose of study drug until 30 days after last dose (Up to 1899 days)
Population: SAF
Measure: Number; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 52
Participants | 36

2. Secondary Outcome: Percentage of Participants With Confirmed Prostate-specific Antigen (PSA) Response
Description: Confirmed PSA response rate was defined as the percentage of participants with >= 50% decline in PSA from baseline to the lowest postbaseline PSA result, with a consecutive assessment conducted at least 3 weeks later to confirm the PSA response.
Time Frame: Baseline (Day 1); Days 29, 57, 85, 169 and then every 84 days until 30 days after the last dose (up to Day 1899)
Population: Full Analysis Set (FAS): The FAS consisted of all participants who received at least one dose of study drug and had at least one post baseline measurement.
Measure: Number; unit: Percentage of Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 50
Percentage of Participants | 46

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days after last dose (Up to 1899 days)
Description: The Safety analysis set (SAF) consisted of all participants who took at least one dose of the study drug.
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 6/52
Serious Adverse Events (participants affected / at risk) | 10/52
Other Adverse Events (participants affected / at risk) | 25/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=52)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide (N=52)
Constipation (Gastrointestinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (4)
Asthenia (General disorders) | 5 (7)
Pain (General disorders) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/60/NCT03641560/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT03641560/SAP_003.pdf